CLINICAL TRIAL: NCT01958814
Title: Controlled Randomized Double-blind Study Comparing Salbutamol and Placebo Via Aerosol in Chronic Obstructive Respiratory Insufficiency in Exacerbartion Treated With Noninvasive Ventilation
Brief Title: Beta Agonist Nebulization in Non Invasively Ventilated COPD Patients: Safety, and Therapeutic Efficacy Range.
Acronym: BANNISTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHAO11-PD / BANNISTER; 2011-004802-20 (EudraCT Number)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2016-05

CONDITIONS: Chronic Respiratory Failure
MeSH Terms: interventions — Albuterol; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salbutamol - Placebo (Experimental): salbutamol at M0 and M60 placebo administration
  Interventions: Drug: Salbutamol; Drug: Placebo
- Placebo - Salbutamol (Experimental): placebo at M0 and M60 salbutamol administration
  Interventions: Drug: Salbutamol; Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — First administration of salbutamol or placebo at M0 and 2nd salbutamol or placebo at M60 (or M0 + 60 minutes)
  Other Names: Treatment
Drug: Placebo — First administration of salbutamol or placebo at M0 and 2nd salbutamol or placebo at M60 (or M0 + 60 minutes)
  Other Names: physiological serum

SUMMARY:
randomized double-blind controlled study in parallel groups

Salbutamol is a β2 mimetic short-acting to be administered by nebulization in this study.

During this administration, non invasive ventilation for the patient will be continued.

DETAILED DESCRIPTION:
Randomization will focus on the treatment administered (placebo or salbutamol ).

After the first phase , a switch will be set up for each patient , retaining the blind it will be administered salbutamol (for those who received placebo in the first phase ) or placebo (for those receiving salbutamol ) .

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with BPCO, defined:

  * by an irreversible obstructive syndrome
  * and\or by different arguments (histories, symptoms, physical examination, thoracic radiography, gas of the blood)
* Decompensation of this BPCO in the form of acute respiratory failure
* No argument for a dominant acute left cardiac insufficiency
* Consent signed by the patient
* Patient with national health assurance

Exclusion Criteria:

* Contraindications in the not invasive ventilation
* Patient not volunteer for the realization of the spirometry
* Precautions for use of ß2 mimetic (engrave hyperthyroidism)
* Under guardianship patient or protection of justice
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Collection at the bedside spirometric values | gross change in forced expiratory volume in one second from the beginning of salbutamol or placebo and 15 min after the start

SECONDARY OUTCOMES:
gross change in vital capacity of peak expiratory flow rate, the ratio of FEV, forced expiratory flow | between the median baseline and 15 min after the start of treatment
gross change in respiratory rate, heart rate and systolic and diastolic blood pressure | between baseline and 15 min after the start of treatment
gross change in dyspnea | between baseline and 15 min after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François DEQUIN, MD-PhD, Principal Investigator — CHRU de TOURS
Locations (3):
- France (3):
  - Service de Réanimation Médicale - CHR d'Orléans, Orléans
  - Service de Réanimation, Poitiers
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bodet-Contentin L, Guillon A, Boulain T, Frat JP, Garot D, Le Pennec D, Vecellio L, Ehrmann S, Giraudeau B, Tavernier E, Dequin PF. Salbutamol Nebulization During Noninvasive Ventilation in Exacerbated Chronic Obstructive Pulmonary Disease Patients: A Randomized Controlled Trial. J Aerosol Med Pulm Drug Deliv. 2019 Jun;32(3):149-155. doi: 10.1089/jamp.2018.1484. Epub 2018 Dec 27. PMID 30589607